CLINICAL TRIAL: NCT05263531
Title: The Safety and Efficacy of Remote Ischemic Conditioning on Motor Recovery After Acute Stroke
Brief Title: Remote Ischemic Conditioning for Motor Recovery After Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor of Neurosurgery, Vice-President of Xuan Wu Hospital, Capital Medical University, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIC-MR
Record Dates: First submitted 2020-12-01; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-08

CONDITIONS: Ischemic Stroke
Keywords: remote ischemic conditioning
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote ischemic conditioning (Experimental): Receiving remote ischemic conditioning (RIC) treatment with pressure set at 200 mmHg.
  Interventions: Device: remote ischemic conditioning
- placebo remote ischemic conditioning (Sham Comparator): Receiving sham RIPC treatment with pressure set at 60 mmHg
  Interventions: Device: remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on bilateral arms and inflated to design pressure for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.

SUMMARY:
The most recent treatment for stroke rehabilitation is to combine physical training with other therapies to enhance or accelerate recovery.The hypothesis of this study is that remote ischemic conditioning (RIC) might have a beneficial effect on motor recovery of AIS

DETAILED DESCRIPTION:
Despite the effective reperfusion therapies ,acute ischemic stroke(AIS) is still one of the leading causes of disability, resulting in an economic burden. Multidisciplinary rehabilitation has benefit effects on motor recovery and remains the first-line intervention strategy for attenuating motor function impairments. However, the effect of the physiotherapy application alone is not satisfactory, The potential treatment effect of RIC on motor recovery of AIS has not been investigated. The investigators designed this randomized clinical trial to examine whether RIC has a beneficial effect on poststroke motor function recovery.There are 2 arms in this trial: One arm is RIC treatment, the other one is sham RIC treatment. The motor function will be assessed by Fugl-Meyer Motor Scale before and after the treatment to evaluate its exact effect on motor recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-80 years;
2. First-ever unilateral ischemic stroke,5~10 days after onset;
3. Had motor dysfunction caused by stroke(Fugl-Meyer≤55)
4. mRS≤1 before stroke
5. NIHSS 6~20
6. Written consent was obtained from the subject.

Exclusion Criteria:

1. Cannot complete assessments-ie, psychiatric disorders, sensory aphasia, dementia
2. brainstem lesion or cerebellun lesion
3. poorly controlled diabetes mellitus
4. Application of agent which thought to impair or improve recovery based on laboratory and clinical evidence within 1 month (ie,DA,MAOI, SSRI,α1/α2 adrenergic receptor inhibitors,BZD,etc)
5. severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
changes in Fugl-Meyer score | 0-3 months
  Fugl-Meyer scale assessment (FMA) will be used for assessing improvement of motor function. Total score of FMA range from 0 to 100, a score of 100 means full recovery of motor function

SECONDARY OUTCOMES:
Changes of the level of angiogenesis related factors | 0-3 months
  circulatory VEGF,EGF,PDGF,CD40L will be tested before and after the treatment
changes in Barthel Index | 0-3months
  Barthel Index will be used for assessing ability of daily life, range from 0 to 100, the higher the score, the better recovery patient reach

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD PhD, Principal Investigator — Capital Medical University Xuan Wu Hospital
Locations (1):
- Xuan Wu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes